CLINICAL TRIAL: NCT04081987
Title: A Multi-center, Prospective, Pilot Study Intended for Data Collection to Evaluate and Calibrate a Novel Non-invasive Wearable Device for Monitoring Vital Signs
Brief Title: Evaluation and Calibration of a Novel Non-invasive Wearable Device for Monitoring Vital Signs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BiPS Medical (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BiPS
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Post-cardiac Surgery; Intensive Care Unit Patients
Keywords: Arterial line; Non-invasive monitoring; Vital signs; Blood pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non-invasive monitoring — Comparing blood pressure (diastolic & systolic), heart and respiration rates, blood oxygen level and body temperature measurement using the BiPS non-invasive monitor to an arterial line.

SUMMARY:
The purpose of this clinical study is to compare the measurement of vital signs (blood pressure, heart rate, respiration rate, blood oxygen levels and body temperature) measured by the non-invasive, continuous and wireless BiPS monitoring device with vital signs measured by current standard of care hospital equipment (blood pressure measurements will be obtained from arterial line) an invasive arterial line. The study will be conducted in two medical centers in Israel and include 50 adult patients that are connected to an arterial line as part of their routine care.

DETAILED DESCRIPTION:
BiPS Medical has developed a wearable, wireless device that conveniently monitors important vital sign trends over time - blood pressure (diastolic & systolic), heart and respiration rates, blood oxygen level (SPO2) and body temperature - to aid in identifying clinical deterioration. The device is base on a combination of inflatable mini finger cuff and photoplethysmograph technology.

The aim of this study is to collect data for evaluating and calibrating of the BiPS monitor for monitoring patient vital signs and compare it to current standard of care hospital monitors. The study population includes a total of 50 adult patients that are connected to an arterial line as part of their routine care. The BiPS non-invasive monitor will be attached to participating patients during their stay in the ICU/ recovery in cardiac ICU/Post Anesthesia Care Unit /other hospital designated unit. The device will be placed on the patient for 60 minutes while in hospital bed, in which up to 20 blood pressure measurements are performed (each takes up to 60 seconds). Heart and respiration rates, body temperature and SPO2 will be measured continuously while the device is attached to the patient hand.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who agree to sign an informed consent.
* Patients connected to an arterial line as part of their routine care (e.g., patients recovering from cardiac or other major surgery)

Exclusion Criteria:

* Pregnant women.
* Patients under the age of 18.
* Patients who are not connected to an arterial line as part of their routine care.
* Unable to give informed consent.
* Patients with poor or no finger pulse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include a total of 50 adult patients that are connected to an arterial line as part of their routine care (e.g., post operative cardiac patients, or intensive care unit patients), recruited in Sourasky Medical Center (Ichilov), Tel-Aviv and Carmel Medical Center, Haifa.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Level of accordance between the BiPS monitor and the arterial line | 60 minutes
  Correlation between the vital sgns measured on The BiPS non-invasive monitor and those measured through the arterial line

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Carmel Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will probably share the experimental results showing the level of accordance between the two measurement methods, but not the information of each participant separately.